CLINICAL TRIAL: NCT02919956
Title: Cerebral Anatomy, Hemodynamics and Metabolism In Single Ventricles: Relationship to Neurodevelopment
Brief Title: Cerebral Anatomy, Hemodynamics and Metabolism
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-012291; 5R01HL090615-09 (NIH)
Record Dates: First submitted 2016-08-02; First posted 2016-09-30 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Single Ventricle; Fontan
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Univentricular Heart | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Group I: CBF-I Single Ventricles: The 1st group (cohort group) will be patients who were enrolled in the original NIH CBF grant. These patients will undergo a 60-90 minute Magnetic Resonance Imaging scan of the brain and heart. They will also have Neurodevelopmental Testing.
  Interventions: Other: Magnetic Resonance Imaging; Other: Neurodevelopmental Testing
- Group II: Prospective Single Ventricles: The 2nd group (cross sectional group) will be prospectively recruited from SV patients after Fontan operation but were not participants in the original study and will be age matched to Group I to enrich the patient population. These patients will undergo a 60-90 minute Magnetic Resonance Imaging scan of the brain and heart. They will also have Neurodevelopmental Testing.
  Interventions: Other: Magnetic Resonance Imaging; Other: Neurodevelopmental Testing
- Group III: CBF-I Normal Controls: The 3rd group (cohort group) will be normal controls who were enrolled in the original CBF grant. These patients will have Neurodevelopmental Testing. The data from these patients' MRI from CBF-I (original CBF grant) will be used.
  Interventions: Other: Neurodevelopmental Testing
- Group IV: Prospective Normal Controls: The 4th group (cross sectional group) will be prospectively recruited from patients who come to Children's Hospital of Philadelphia (CHOP) for clinically indicated MRIs and found to have structurally normal cardiac and brain anatomy. These patients will have an abbreviated research MRI, lasting 15-20 minutes, added onto their clinically-indicated MRI at CHOP. They will also have Neurodevelopmental Testing.
  Interventions: Other: Magnetic Resonance Imaging; Other: Neurodevelopmental Testing
- Volunteer Group: There will also be a volunteer group of one to five volunteers that will be enrolled prior to enrollment in the other four study groups. These volunteers will be prospectively recruited from patients who come to Children's Hospital of Philadelphia (CHOP) for a clinically-indicated MRI and consent to have an additional 15-20 minutes of research MRI scanning. The purpose will be to ensure that the brain MRI sequences run correctly and produce useful information before the patient and normal control enrollment begins. The volunteers will not undergo neurodevelopmental testing.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — An MRI scan takes pictures of the brain and heart using a magnet and radio waves. During scanning, measurements of oxygen delivery to the brain will be obtained (CMRO2) as well as evaluation of the heart as it relates to the brain. During the scan patients will be monitored for safety by ECG, blood pressure, television camera, pulse oximetry, and carbon dioxide measurements. Cardiac anesthesiologist and cardiologist will be present.
  Other Names: MRI
  Groups: Group I: CBF-I Single Ventricles; Group II: Prospective Single Ventricles; Group IV: Prospective Normal Controls; Volunteer Group
Other: Neurodevelopmental Testing — Quantitative ND tests and standardized rating scales will be used in the areas of intellectual, adaptive, visual motor skills, academic achievement in math and reading, attention and executive functioning , motor skills, memory, language, social skills and behavior. Neurodevelopmental Testing will last approximately 3.5-4 hours. Testing will be done through the Neurobehavioral Core at CHOP. Breaks will be taken as needed and a one hour lunch break will be taken, if applicable. ND testing will be performed prior to MRI (if on the same day) or on a different day than the MRI to promote engagement and best performance.
  Other Names: ND Testing
  Groups: Group I: CBF-I Single Ventricles; Group II: Prospective Single Ventricles; Group III: CBF-I Normal Controls; Group IV: Prospective Normal Controls

SUMMARY:
Single ventricle lesions are the leading cause of illness and death from congenital heart disease. The modified Fontan Operation is the corrective surgery for these lesions. The operation is done in stages over a few years and children who complete the operation are known to have greater neurodevelopmental (ND) deficits than the general population. The purpose of this study is to understand how blood flow to the brain (CBF) and brain lesions relate to ND outcome, as well as how CMRO2 relates to anatomic brain lesions. These relationships will be studied through Magnetic Resonance Imaging (MRI) and ND Testing.

DETAILED DESCRIPTION:
Single ventricle (SV) lesions are the leading cause of morbidity and mortality from congenital heart disease (CHD) in the United States. The definitive palliative surgery is the modified Fontan operation where systemic venous return is routed directly to the pulmonary arteries. The surgical reconstruction is performed in stages over a few years which includes the "Stage I" and hemiFontan or bidirectional Glenn operations. These children are known to have greater neurodevelopmental (ND) deficits than the general population and other forms of CHD. For example, a study at Children's Hospital of Philadelphia revealed that at 9 years old, 1/3 were receiving some form of special education; the median intelligence quotient (IQ) was 86 with mental retardation in 18%. One component to ultimate ND outcome is cerebral blood flow (CBF). Preliminary data in SV in the literature across all age ranges and multiple disease states, suggests that CBF is related to ND; a recent review of 25 studies bears this out. Another component to ND outcome is anatomic brain lesions. Preliminary data from a current NIH study of CBF study suggests a link between CBF and brain lesions (decreased CBF is associated with more brain lesions), weaving a complex interaction leading to ultimate ND outcome. There is a pressing need to understand CBF and brain lesions as it relates to childhood ND; this rapid growth stage may be especially important to ultimate cognitive function having not only a humanistic/social impact but a large economic one as well.

Data from a previous NIH grant which ended November 2014 indicates that CBF in SV patients changes throughout the staged surgeries and in the first 2 stages, under stressed conditions such as hypercarbia; in addition, initial look at the data suggests a difference in brain abnormalities as well. These children are especially at risk for altered CBF and brain abnormalities with their changing physiology. At Stage I, a "runoff" physiology is present created by the aorto-pulmonary shunt potentially causing a "steal" from the cerebral circulation. In the 2nd stage (e.g. hemiFontan), cerebral and pulmonary circulations are connected directly and exclusively in series with each other; aortic blood flows to the brain and then directly to the lungs via the superior vena cava. After Fontan completion, downstream cerebral venous pressures are elevated. Finally, SV patients develop aorto-pulmonary collaterals (APC) at all stages and another ongoing research project found a strong inverse correlation between CBF and the degree of APC flow, further putting CBF of SV at risk.

In another study, magnetic resonance imaging (MRI) was utilized to measure blood flow and visualize cerebral anatomy by phase contrast MRI arterial spin labeling and anatomic imaging such as T1 weighted sequences and diffusion tensor imaging. MRI utilizing susceptometry (oximetry) recently developed by an investigator on this renewal, can also quantify the cerebral metabolic rate of oxygen consumption (CMRO2). This combination of MRI capabilities offers a unique opportunity to assess cerebral anatomy, hemodynamics and oxygen metabolism in the same study; by combining this with ND testing, this study is poised to link the two in the hopes of not only understanding cognitive function but to positively intervene in ND outcome. A comprehensive assessment of brain anatomy and function linked to ND outcomes has never been reported in any group of patients nor with utilizing measures at 2 time points.

This is a prospective, single center study of SV patients and seeks to relate cerebral anatomy, hemodynamics and CMRO2 with ND outcome using another patient cohort obtained under a previous study as a basis and utilizing data from 2 time points (original grant and renewal). This approach along with using cerebral carbon dioxide (CO2) reactivity and CMRO2 are major strengths of this study. Elucidating these factors may ultimately lead to modifications in management (e.g. timing of surgery) and identifying children at cognitive risk to implement early intervention and possibly improve ND outcome.

ELIGIBILITY:
Inclusion Criteria:

SV Patients

* Subjects ages 3 to 15 years old who have completed their Fontan procedure and their parents/guardians.
* Any complex congenital heart lesion that has SV physiology of either right ventricle (RV) or left ventricle (LV) morphology.
* Ability to undergo a 60-90 minute MRI scan under general anesthesia or deep sedation if general anesthesia or sedation is needed.
* Parents signing informed consent. Healthy Controls
* Males and females ages 3 to 15 years old if in the original cohort and if not in the original cohort, age matched with Groups I and II, and their parents/guardians.
* Normal cerebral and cardiac anatomy who are normocephalic and who are asymptomatic.
* For normal controls being prospectively enrolled and not part of the original grant, the ability to extend the clinical MRI an extra 15-20 minutes.
* For normal controls undergoing sedation, the ability to extend anesthesia for approximately 15-30 minutes for research purposes only.
* Parents signing informed consent. Volunteers
* Patients who come to CHOP for a clinically indicated MRI.
* The ability to extend the clinical MRI an extra 15-20 minutes.
* If 18 or over, patient signing informed consent.
* If under 18, parents signing informed consent.

Exclusion Criteria:

SV Patients

* A patient whose primary language is not English. Patients who speak English who have parents or guardians who do not speak English would not be excluded.
* Any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any known significant neurological disease outside of the usual state of SV patients.
* Any major anomalies which would confound neurological outcome.
* A patient with a pacemaker or cardioverter/defibrillator in place.
* A contraindicated ferromagnetic foreign body).
* Pregnancy Healthy Controls
* An individual whose primary language is not English. Patients who speak English who have parents or guardians who do not speak English would not be excluded
* Any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any known significant neurological disease.
* Any contraindication to extending the MRI.
* Pregnancy. Volunteers
* A patient whose primary language is not English. Patients who speak English who have parents or guardians who do not speak English would not be excluded.
* Any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contraindication to extending the MRI.
* Pregnancy.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group I (cohort) will be patients enrolled in the original NIH CBF grant. Group II (cross-sectional) will be recruited from SV patients after Fontan operation but were not participants in the original study to enrich the patient population and to maximize Group I enrollment. Group III will be normal controls enrolled in the original CBF grant. Group IV will be patients at The Children's Hospital of Philadelphia (CHOP) for clinical MRIs and found to have structurally normal cardiac and brain anatomy. Parents/guardians of Group I-IV patients will be enrolled, as well. There will be a group of 1-5 volunteers enrolled to test the study MRI protocol. Volunteers will be patients who come to CHOP for clinical MRIs.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-04; Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Relationship of CBF and Brain Abnormalities to ND Outcomes | Up to 10 years
  This study proposes to recall SV patients from a cohort from a previous study to undergo an MRI (for anatomy, CBF and CMRO2) and ND testing. Normals from a previous grant will also be recalled to undergo ND testing. Correlations will be performed between ND, CBF and brain abnormalities from the a) original MRI, b) current study and c) change between the two. Response to hypercarbia will be assessed in a select group of patients. Additional SV patients and normals will be recruited to enrich the population. In addition, this study will determine how CBF and brain abnormalities in SV patients evolve over the course of time. Therefore, the timeframe for the comparisons will be a) from the original MRI to the current MRI and neurodevelopmental testing (up to 10 years) as well as b) the current MRI with neurodevelopmental testing.

SECONDARY OUTCOMES:
Relationship of CMRO2 to ND outcome | Up to 10 years
  This Aim will correlate CMRO2 as assessed in MRIs performed in the current study from Aim 1 to ND outcome. In addition, this proposal will relate CMRO2 to anatomic brain lesions by MRI. Therefore, the timeframe for the comparisons will be a) from the original MRI to the current MRI and neurodevelopmental testing (up to 10 years) as well as b) the current MRI with neurodevelopmental testing.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Fogel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Felix Werhil from the University of Penn will be analyzing the CMRO2 studies from the MRI images. Data will be transferred to him on a flash drive that has been encrypted and password-protected according to CHOP IT standards and hand delivered by the PI or a member of the study team.
  Dr. Alexandra Hanlon from University of Penn School of Nursing will be performing the statistics for the study. Investigators will have a REDCap database, which Dr. Hanlon has been approved for and received CHOP identity to access.

REFERENCES:
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Norwood WI, Kirklin JK, Sanders SP. Hypoplastic left heart syndrome: experience with palliative surgery. Am J Cardiol. 1980 Jan;45(1):87-91. doi: 10.1016/0002-9149(80)90224-6. PMID 6153137
- [Background] Norwood WI, Lang P, Hansen DD. Physiologic repair of aortic atresia-hypoplastic left heart syndrome. N Engl J Med. 1983 Jan 6;308(1):23-6. doi: 10.1056/NEJM198301063080106. No abstract available. PMID 6847920
- [Background] Seliem M, Muster AJ, Paul MH, Benson DW Jr. Relation between preoperative left ventricular muscle mass and outcome of the Fontan procedure in patients with tricuspid atresia. J Am Coll Cardiol. 1989 Sep;14(3):750-5. doi: 10.1016/0735-1097(89)90121-6. PMID 2527902
- [Background] Whitehead KK, Gillespie MJ, Harris MA, Fogel MA, Rome JJ. Noninvasive quantification of systemic-to-pulmonary collateral flow: a major source of inefficiency in patients with superior cavopulmonary connections. Circ Cardiovasc Imaging. 2009 Sep;2(5):405-11. doi: 10.1161/CIRCIMAGING.108.832113. Epub 2009 Jul 8. PMID 19808629
- [Background] Glatz AC, Rome JJ, Small AJ, Gillespie MJ, Dori Y, Harris MA, Keller MS, Fogel MA, Whitehead KK. Systemic-to-pulmonary collateral flow, as measured by cardiac magnetic resonance imaging, is associated with acute post-Fontan clinical outcomes. Circ Cardiovasc Imaging. 2012 Mar;5(2):218-25. doi: 10.1161/CIRCIMAGING.111.966986. Epub 2012 Jan 6. PMID 22228054
- [Background] Dori Y, Glatz AC, Hanna BD, Gillespie MJ, Harris MA, Keller MS, Fogel MA, Rome JJ, Whitehead KK. Acute effects of embolizing systemic-to-pulmonary arterial collaterals on blood flow in patients with superior cavopulmonary connections: a pilot study. Circ Cardiovasc Interv. 2013 Feb;6(1):101-6. doi: 10.1161/CIRCINTERVENTIONS.112.972265. Epub 2013 Jan 15. PMID 23322742
- [Background] Grosse-Wortmann L, Al-Otay A, Yoo SJ. Aortopulmonary collaterals after bidirectional cavopulmonary connection or Fontan completion: quantification with MRI. Circ Cardiovasc Imaging. 2009 May;2(3):219-25. doi: 10.1161/CIRCIMAGING.108.834192. Epub 2009 Mar 25. PMID 19808596
- [Background] Mahle WT, Tavani F, Zimmerman RA, Nicolson SC, Galli KK, Gaynor JW, Clancy RR, Montenegro LM, Spray TL, Chiavacci RM, Wernovsky G, Kurth CD. An MRI study of neurological injury before and after congenital heart surgery. Circulation. 2002 Sep 24;106(12 Suppl 1):I109-14. PMID 12354718
- [Background] Fontan F, Baudet E. Surgical repair of tricuspid atresia. Thorax. 1971 May;26(3):240-8. doi: 10.1136/thx.26.3.240. PMID 5089489
- [Derived] Fogel MA, Donnelly E, Crandell I, Hanlon A, Whitehead KK, Harris M, Partington S, Biko D, Flynn T, Nicolson S, Gaynor JW, Licht D, Vossough A. Cerebral Blood Flow, Brain Injury, and Aortic-Pulmonary Collateral Flow After the Fontan Operation. Am J Cardiol. 2023 Dec 1;208:164-170. doi: 10.1016/j.amjcard.2023.08.023. Epub 2023 Oct 14. PMID 37844519